CLINICAL TRIAL: NCT03705611
Title: Secondary Distribution of HIV Self-tests Through Antenatal and HIV Testing Services: a Pragmatic Cluster-randomized Trial (STAR-ANC)
Brief Title: Secondary Distribution of HIV Self-tests Through Antenatal Care Clinic Attendees and Index Clients
Acronym: ANC/FRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: World Health Organization (Other); Liverpool School of Tropical Medicine (Other); UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14916
Record Dates: First submitted 2018-06-01; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-05

CONDITIONS: HIV/AIDS; HIV Infections
Keywords: Secondary distribution; HIV self-testing; Malawi
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Intervention Model Description: 1:1:1 randomization of primary health clinics (cluster randomized trial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (No Intervention): Provide personalised clinic invitation slips (letters) to partners to come for HIV testing, and to access post-test services
- HIV self-testing only (Experimental): HIV self-testing only
  Interventions: Diagnostic Test: HIV self-testing only
- HIV self-testing secondary accuracy (Experimental): HIV self-testing secondary accuracy
  Interventions: Diagnostic Test: HIV self-testing only; Behavioral: HIV self-testing secondary accuracy

INTERVENTIONS:
Diagnostic Test: HIV self-testing only — Partners will be asked to self-test for HIV following receipt of the test kit from their sexual contact at home or in the community. They will also get information about the partner's clinic -- an HIV testing service room dedicated to providing HIV testing, confirmatory HIV testing, and referral to HIV treatment and prevention services including couples counselling.
  Other Names: OraQuick, OraSure Technologies, USA
  Arms: HIV self-testing only; HIV self-testing secondary accuracy
Behavioral: HIV self-testing secondary accuracy — A monetary incentive provided conditional on clinic attendance and fulfillment of secondary accuracy procedures such as undergoing on spot finger prick rapid HIV testing
  Arms: HIV self-testing secondary accuracy

SUMMARY:
A three arm cluster randomized trial randomizing government primary health clinics to a) standard of care (SOC) with clinic invitation only; b) standard of care (SOC) and one self-test kit to give to sexual partner (s); c) standard of care (SOC) and self-test kit and monetary incentive given to partner conditional on clinic attendance and completion of pre-set procedures to determine secondary accuracy.

Trial to be conducted in four districts (Blantyre, Zomba, Machinga and Chikwawa) in Malawi in collaboration with the Ministry of Health.

Two primary outcomes:

1. proportion of male partners of antenatal care clinic attendees reported by the woman to have tested for human immunodeficiency virus (HIV) within 28 days of enrolling the woman
2. Number of new HIV positives identified by providing trial services to newly tested HIV positive clients in routine HIV testing service within 28 days of enrolling the index client.

Data analysed as intention to treat with all eligible antenatal care (ANC) attendees and index clients at each health facility as the denominator, with unpaired t-test used to compare each intervention arm to the standard of care (SOC).

DETAILED DESCRIPTION:
Type of study: This proposal is for a 3-arm pragmatic cluster randomised trial (CRT) using primary care clinics as the unit of randomisation. The three arms are: 1) Standard of care (SOC) with written invitation to the partner, and two intervention arms of 2) standard of care (SOC) + HIV self-test kits delivered by the partner; and 3) arm 2 plus a monetary incentive for partners who participate in a linked-accuracy study.

Problem: Malawi's Ministry of Health (MoH) uses a highly decentralized approach for delivery of HIV services that delivers over 3 million HIV tests each year, and has taken the country close to The Joint United Nations Programme on HIV and AIDS (UNAIDS) 90-90-90 targets. However, a testing gap remains among populations with barriers to accessing facility-based HIV testing services (HTS), including men. The investigators recently showed partner-delivered (secondary distribution) of HIV self-testing (HIVST) kits, via women attending antenatal care (ANC) in urban Blantyre, to be effective at increasing the uptake of HIV testing and subsequent HIV care and prevention services among male partners. However, unanswered questions that remain to be addressed include:

* the accuracy of HIV self-testing (HIVST) when kits are provided by secondary distribution
* how effective secondary distribution is when fully devolved to Ministry of Health (MoH) providers ("pragmatic")
* whether the high safety profile and acceptability of secondary distribution of HIV self-test kits from antenatal care (ANC) clinics can be generalised to other clinic services.

Role of Ministry of Health (MoH), implementers and researchers: HIV self-test kits will be delivered by the HIV Department of Ministry of Health (MoH), Malawi, in partnership with Population Services International (PSI)-Malawi. Ministry of Health (MoH) aims to routinely scale-up secondary distribution from antenatal care (ANC) clinics in high HIV prevalence districts, and HIV testing services (HTS) nationally if results are satisfactory.

Research Question: Can secondary distribution of HIV self-tests through antenatal care and HIV testing services improve coverage of HIV testing in sexual partners of pregnant women and newly-diagnosed people living with HIV (PLHIV), while maintaining low costs and acceptable linkage, safety and accuracy?

Objectives: The broad objective is to determine the feasibility, benefits, costs, safety and accuracy of secondary distribution of HIV self-test kits from routine antenatal and HIV testing services (HTS) clinics in Malawi. The specific aims are to conduct a pragmatic cluster randomized trial to:

1. Assess the feasibility of programmatic implementation of secondary distribution of HIV self-test kits from routine Ministry of Health (MoH) clinics.
2. Establish the effectiveness of secondary distribution of HIV self-test kits on:

   1. HIV testing among male partners of antenatal care (ANC) attendees
   2. Initiation of antiretroviral therapy (ART) and uptake of voluntary medical male circumcision (VMMC) among male partners of antenatal care attendees
   3. Disclosure and couple testing among male partners of antenatal care attendees
   4. Identification of HIV-positive contacts among partners of newly diagnosed HIV-positive index clients through routine HIV testing services (HTS).
3. Investigate the impact of secondary distribution of HIV self-test kits on the frequency of social harms affecting distributors of HIV self-test kits
4. Estimate the costs and cost-effectiveness of adding secondary distribution of HIV self-test kits to the antenatal care and HIV testing service.
5. Estimate the sensitivity and specificity of OraQuick HIV self-test kits under secondary distribution.

Methodology Participants and intervention Pregnant women registering for antenatal care in 27 primary health clinics and newly diagnosed HIV+ clients from the same 27 clinics in Blantyre, Chikwawa, Machinga and Zomba Districts. Restricted randomisation will be used to allocate clinics to the 3 arms (1:1:1). Ministry of Health (MoH) Clinic staff in the HIV self-testing arms will be trained in use of oral HIVST kits (OraQuick). HIV self-test kit supply will use Ministry of Health (MoH) supply chains. Information and educational materials will include a tablet with a video clip demonstrating correct use of kits. Data capture tools and training materials will be developed with Ministry of Health (MoH).

A full-time research assistant will support research-data capture at each clinic. For the accuracy sub-study this will include a brief questionnaire, repeat HIV testing (2 finger-prick HIV rapid diagnostic tests plus repeat OraQuick) and dried blood spots (DBS) for antiretroviral therapy (ART) drug and HIV viral load testing.

Primary and secondary outcomes:

The two primary outcomes are comparison between standard of care (SOC) and HIV self-testing arms of:

1. % of women reporting that their partner has tested for HIV within 28 days of ANC appointment.
2. Number of previously undiagnosed people living with HIV (PLHIV) identified among partners of HIV-positive index patients by Day 28

The six secondary outcomes are:

1. % of partners of antenatal care attendees who start antiretroviral therapy (ART), undergo voluntary medical male circumcision (VMMC), or attend discordant couples clinic within 28 days of enrolling the woman
2. % of partners of antenatal care attendees who attend the clinic for any HIV services within 28 days of enrolling the woman
3. % HIV+ index clients who self-report at least one partner tested for HIV as a result of their diagnosis, measured at Day 28
4. Number of partners of HIV testing services (HTS) index clients who start antiretroviral therapy (ART), or undergo voluntary medical male circumcision (VMMC), or attend discordant couples clinic within 28 days of index diagnosis
5. Number of partners of HIV+ Index clients who attend the clinic for any HIV services within 28 days of index diagnosis
6. Risk of adverse events (e.g. partnership breakdown, intimate partner violence, etc.) related to self-testing reported by antenatal care / HIV-positive index clients, measured at Day 28

Sample size:

9 clinics per arm each recruiting 350 antenatal care clients and 135 newly diagnosed people living with HIV (PLHIV) will provide 90% power to detect a 12% absolute difference in the primary outcome, assuming 20% of standard of care (SOC) partners, and a coefficient of variation (k) of 0.25. Cluster-level summaries with a t-test applied to the mean of clinic proportions will be compared to the standard of care (SOC) for the primary outcome.

Ethical considerations: The investigators request a waiver of informed consent for HIV self-testing, as this is now international best practice, and delivery will be by Ministry of Health (MoH) routine systems. Written informed consent (witnessed thumb-print if illiterate) will be taken from all participants in the accuracy sub-study.

Dissemination: The results will be used to inform Ministry of Health (MoH) on HIV self-testing scale-up plans, and will also be disseminated through College of Medicine in Blantyre including College of Medicine Research Ethics Committee (COMREC), and through conference presentations and publication in peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria for clinics (cluster):

* Government primary health clinic or centre
* Provides antenatal care services, HIV testing services and HIV treatment services

Exclusion Criteria for clinics:

* Not a government health facility
* Does not provide antenatal care services, HIV testing services and HIV treatment services
* Not willing to be part of the trial

Individual level eligibility screen for antenatal care attendees:

* First antenatal care visit
* Age 18 years or older
* Has one main sexual partner (i.e. likely father)
* Main sexual partner not already known to be HIV-positive and on antiretroviral therapy
* Sexual partner likely to remain in clinic catchment area for the next 28 days
* Not already tested together in this pregnancy [e.g. partner has come with her on this visit and has tested today]
* Not already recruited in the study

Individual level eligibility screen for index clients:

* Age 18 years or older
* At least one sexual partner not already known to be HIV-positive and on antiretroviral therapy
* At least one sexual partner likely to remain in catchment area within the next 28 days
* Not already recruited in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of partners tested for HIV | 28 days
  For antenatal care clinic attendees, this is as reported by the women during their next antenatal care visit
Number of newly diagnosed HIV positive people | 28 days
  A count of number of sexual contacts of index HIV positive clients attending the clinic for post-test services

SECONDARY OUTCOMES:
Proportion of partners of antenatal care clinic attendees who start HIV treatment, undergo circumcision, or attend discordant couples clinic | 28 days
Risk of adverse events (e.g. partnership breakdown, intimate partner violence, etc.) related to self-testing reported by antenatal care clinic attendees or HIV-positive index clients | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Desmond, PhD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Mulanje District Hopsital, Mulanje, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data relating to the primary and secondary outcomes will be made publicly available through the London School of Hygiene & Tropical Medicine Data Campus
Supporting Information: Study Protocol, SAP
Time Frame: After the main results have been published
Access Criteria: Contact the principal investigator for authorization to re-use the data
URL: http://datacompass.lshtm.ac.uk/

REFERENCES:
- [Derived] Choko AT, Fielding K, Johnson CC, Kumwenda MK, Chilongosi R, Baggaley RC, Nyirenda R, Sande LA, Desmond N, Hatzold K, Neuman M, Corbett EL. Partner-delivered HIV self-test kits with and without financial incentives in antenatal care and index patients with HIV in Malawi: a three-arm, cluster-randomised controlled trial. Lancet Glob Health. 2021 Jul;9(7):e977-e988. doi: 10.1016/S2214-109X(21)00175-3. PMID 34143996